CLINICAL TRIAL: NCT06575751
Title: Cannabidiol and Cannabis Concentrate Users: A Randomized, Placebo Controlled Study
Brief Title: Cannabidiol and Cannabis Concentrate Users
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-0953; 1P50DA056408 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blind to medication assignment, as will all care providers and investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Broad Spectrum Cannabidiol (bsCBD) 400 mg (Active Comparator): bsCBD in a 400 mg dose will be used as described in the study arms.
  Interventions: Drug: Broad Spectrum Cannabidiol (bsCBD) 400 mg
- Broad Spectrum Cannabidiol (bsCBD) 200 mg (Active Comparator): bsCBD in a 200 mg dose will be used as described in the study arms.
  Interventions: Drug: Broad Spectrum Cannabidiol (bsCBD) 200 mg
- Placebo (Placebo Comparator): A medically inert placebo medication will be used as described in the study arms.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Broad Spectrum Cannabidiol (bsCBD) 400 mg — Participants in this Arm will take 400 mg of bsCBD daily. Participants will take medication by mouth with food in the morning and evening.
  Arms: Broad Spectrum Cannabidiol (bsCBD) 400 mg
Drug: Broad Spectrum Cannabidiol (bsCBD) 200 mg — Participants in this Arm will take 200 mg of bsCBD daily. Participants will take medication by mouth with food in the morning and evening.
  Arms: Broad Spectrum Cannabidiol (bsCBD) 200 mg
Drug: Placebo — Participants in this Arm will take a medically inert placebo. Participants will take medication by mouth with food in the morning and evening.
  Arms: Placebo

SUMMARY:
This study is a randomized, placebo-controlled, dose-ranging trial of plant-derived cannabidiol (CBD) among people who regularly use cannabis concentrates but are not trying to stop or cut down on their use. The main questions it aims to answer are whether CBD, relative to placebo, reduces cannabis concentrate use, the subjective effects of cannabis, or cannabis craving. Participants will take CBD (200 mg or 400 mg per day) or placebo for 4 weeks and will complete three visits during the study medication period, all conducted using a mobile laboratory.

DETAILED DESCRIPTION:
The overarching aim of this proposal is to combine a naturalistic cannabis administration paradigm with a placebo-controlled, dose-ranging randomized controlled trial of plant-derived cannabidiol (CBD) to evaluate CBD effects on cannabis concentrate use, subjective effects, and cannabis cue reactivity. To achieve this aim, 120 adult frequent concentrate users will be recruited to complete a four-week protocol during which they will complete three sessions in a mobile pharmacology laboratory. Up to 200 participants may be consented/enrolled to account for screen failures and attrition. In two of the sessions, participants will use their typical cannabis concentrate on an ad libitum basis. Amount of delta-9-tetrahydrocannabinol (THC) self-administration during these sessions will be quantified by THC blood levels, obtained in the mobile lab immediately before and after use. Subjective drug effects and exogenous and endogenous cannabinoid biomarkers will also be quantified before and after THC use. Immediately after the first mobile lab session, participants will be randomly assigned to take either 200 mg or 400 mg of plant-derived, broad-spectrum CBD or matched placebo (40 participants per group) daily for four weeks. Participants will complete a second mobile lab session after two weeks to provide a blood sample that will be analyzed for cannabinoid levels. At this session, participants will also complete a cannabis cue reactivity paradigm. Participants will complete a second mobile lab session after four weeks of study medication ingestion, during which blood draws and THC self-administration will be repeated.

There are three aims:

Aim 1. Test the effect of CBD, relative to placebo and to baseline, on cannabis use over four weeks and THC self-administration in the mobile laboratory.

Hypothesis 1a. Both doses of CBD, relative to placebo, will reduce THC metabolite levels at weeks 2 and 4.

Hypothesis 1b. Both doses of CBD, relative to placebo and to baseline, will reduce the amount of THC that participants choose to consume in the mobile laboratory, as assessed by pre- vs. post-use THC blood levels.

Aim 2. Test the effect of CBD, relative to placebo and to baseline, on subjective drug effects (intoxication, psychotomimetic symptoms, anxiety, and negative affect) following acute cannabis concentrate use.

Hypothesis 2. Both doses of CBD, relative to placebo and to baseline, will reduce intoxication, paranoia, anxiety, and negative affect following acute use, even after controlling for between-group differences in amount of concentrate used.

Aim 3. Test the effect of CBD, relative to placebo, on cannabis cue-elicited craving and evaluate whether this effect mediates CBD effects on cannabis use.

Hypothesis 3a. Both doses of CBD, relative to placebo, will reduce cannabis craving.

Hypothesis 3b. CBD's effect on craving at week 2 will mediate its effect on THC metabolite levels at week 4.

For all aims, a linear effect of CBD dose is hypothesized, with the greatest effects in the 400 mg CBD group. Successful achievement of these aims will allow determination of an efficacious dose of CBD that reduces high-THC cannabis use, subjective drug effects, and craving, setting the stage for a subsequent RCT of plant-derived CBD to treat these outcomes in treatment-seeking high-THC cannabis concentrate users.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-60.
2. Regular use (at least 4 times per week) of cannabis concentrates for the last year.
3. Not currently seeking to cut down or stop cannabis use.
4. At least one episode of 3 consecutive days of cannabis abstinence with no experience of severe withdrawal symptoms (i.e., >=4 DSM-5 Cannabis Withdrawal symptoms rated as "severe"), in the last 90 days.
5. At least two symptoms of a DSM-5 cannabis use disorder.

Exclusion Criteria:

1. Use of any illicit substance besides alcohol, nicotine, or cannabis (e.g., cocaine, opiates, methamphetamine, MDMA, benzodiazepines, or barbiturates) in the past 60 days, as indicated by self-report and urine toxicology screening at the beginning of each study visit.
2. Use of CBD-containing products other than cannabis concentrates in the past 90 days.
3. Alcohol use on 3 or more days per week, and/or > 3 drinks per drinking day in the past 60 days. Participants must also have a breath alcohol level of 0 at the beginning of each study visit.
4. Daily nicotine use.
5. Meets DSM-5 diagnostic criteria for a psychotic disorder (e.g., schizophrenia, schizophreniform disorder, schizoaffective disorder), bipolar disorder, or major depression with suicidal ideation, or has a history of treatment for these disorders.
6. Current cardiovascular or respiratory disease (e.g., coronary artery disease, severe asthma, chronic obstructive pulmonary disease, etc.)
7. Current use of any psychotropic (e.g., antidepressants, anxiogenics) or hepatotoxic medications.
8. Currently use of anti-epileptic medications (e.g., clobazam, sodium valproate) or medications known to have major interactions with Epidiolex (buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, and/or teriflunomide) or a history of seizures.
9. Current use of strong or moderate CYP3A4 inhibitors or inducers (commonly used examples not captured by other exclusion criteria include protease inhibitors, macrolide antibiotics [e.g., erythromycin], azole antifungals [e.g., ketoconazole], verapamil, and grapefruit juice).
10. Current use of strong or moderate CYP2C19 inhibitors or inducers (commonly used examples not captured by other exclusion criteria include proton pump inhibitors, prednisone, and norethisterone).
11. Current or past hepatocellular disease, as indicated by medical history or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of the normal range at screening.
12. For female participants, pregnancy or trying to become pregnant. A positive pregnancy test at the beginning of any study visit will result in exclusion from ongoing study participation.
13. For female participants, currently lactating.
14. For female patients of childbearing potential, not willing to use at least an approved method of birth control while taking the study medication, unless she is surgically sterile, partner is surgically sterile or she is postmenopausal (one year).
15. Current suicidality risk as indicated during the conduct of the C-SSRS with concurrence after a study physician's or PI evaluation if the response to C-SSRS questions 1 or 2 is "yes".

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in blood 11-Nor-9-carboxy-THC (THC-COOH) levels | 4 weeks
  THC-COOH levels in blood samples collected at baseline, Week 2, and Week 4 of medication ingestion
Difference in blood delta-9-tetrahydrocannabinol (THC) levels | 4 weeks
  THC levels in blood samples collected before and after cannabis use at baseline and at Week 4 of medication ingestion
Difference in cannabis use | 4 weeks
  Total number of days of cannabis use during the 4-week medication period as reported on daily diaries

SECONDARY OUTCOMES:
Difference in cannabis-induced intoxication | 4 weeks
  Drug Effects Questionnaire score following cannabis use at baseline and at Week 4 of medication ingestion (minimum = 0, maximum = 5, higher scores = greater intoxication)
Difference in cannabis-induced subjective effects | 4 weeks
  Addiction Research Center Inventory Marijuana score following cannabis use at baseline and at Week 4 of medication ingestion (minimum = 0, maximum = 12, higher scores = greater subjective effects)
Difference in cannabis-induced psychotomimetic symptoms | 4 weeks
  Psychotomimetic States Inventory paranoia and cognitive disorganization item scores following cannabis use at baseline and at Week 4 of medication ingestion (minimum = 0, maximum = 54, higher scores = greater psychotomimetic symptoms)
Difference in cannabis-induced anxiety and negative affect | 4 weeks
  Profile of Mood States short form tension, vigor, and elation subscale item scores following cannabis use at baseline and at Week 4 of medication ingestion (minimum = 0, maximum = 60, higher scores = greater anxiety and negative affect)
Difference in cannabis craving | 2 weeks
  Marijuana Craving Questionnaire-Short Form score before and after the cannabis cue reactivity procedure at Week 2 of medication ingestion (minimum = 12, maximum = 84, higher scores = greater craving)

OTHER OUTCOMES:
Difference in blood cannabidiol (CBD) levels | 4 weeks
  CBD levels in blood samples collected at baseline, Week 2, and Week 4 of medication ingestion
Adverse effects | 4 weeks
  Adverse effects reported at baseline and Week 4 of medication ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Schacht, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared through a NIDA P50 data sharing resource.